CLINICAL TRIAL: NCT04857424
Title: A Comparative Quality of Life Assessment Between Internal Endoscopic Versus Percutaneous Drainage of Benign and Malignant Biliary Obstruction
Brief Title: Quality of Life Assessment Between Internal Endoscopic Versus Percutaneous Drainage in Biliary Obstruction
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jad P. AbiMansour, Principal Investigator, Mayo Clinic
Other Study IDs: 21-000142
Record Dates: First submitted 2021-04-21; First posted 2021-04-23 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Biliary Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERCP: Subjects with benign and malignant biliary obstruction who have or will undergo endoscopic retrograde cholangiopancreatography (ERCP)
- PTBD: Subjects with benign and malignant biliary obstruction who have or will undergo percutaneous trans-hepatic biliary drainage (PTBD).

SUMMARY:
The aim of this study is to compare the quality of life in subjects with benign and malignant biliary obstruction who have or will undergo endoscopic retrograde cholangiopancreatography (ERCP) and/or percutaneous trans-hepatic biliary drainage (PTBD).

ELIGIBILITY:
Inclusion Criteria:

* Patients with benign biliary obstruction
* Patients with malignant biliary obstruction
* Patients undergoing ERCP and/or PTBD

Exclusion Criteria:

* Patients with gallstone disease
* Patients who will undergo ERCP who have previously underwent a PTBD
* Patients who will undergo PTBD who have previously underwent an ERCP
* Female patients who are pregnant
* Prisoners and other vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 or over with a diagnosis of benign or malignant biliary obstruction who have underwent an ERCP and/or PTBD will be identified through Best Practices Advisory (BPA), referrals from the clinics of GI consultants and the gastroenterology department procedure schedules at Mayo Clinic, Rochester.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in European Quality of Life-5 Dimensions questionnaire score | Baseline, 1 month, 3 months
  Measured using the European Quality of Life-5 Dimensions questionnaire that measures mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The Euro-QOL-5D score is derived from adding the scores from each of the five items. The best possible score is five (i.e., asymptomatic in each item) and the worst possible score is 15 (incapacitated in each item).

CONTACTS AND LOCATIONS:
Overall Officials: Jad AbiMansour, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://clinicaltrials.gov/